CLINICAL TRIAL: NCT01632501
Title: Safety and Efficacy of the Percutaneous Intervention Performed With Devices of a Single-brand
Acronym: Tsunami
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Sao Lucas da PUCRS (Other)
Responsible Party: Principal Investigator, Denise Oliveira, Principal Investigator, Assistent Cardiologist, Hospital Sao Lucas da PUCRS
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCR1TS
Record Dates: First submitted 2012-06-26; First posted 2012-07-03 (Estimated); Last update posted 2012-07-04 (Estimated); Status verified 2011-01

CONDITIONS: Atherosclerotic Heart Disease; Coronary Heart Disease
MeSH Terms: conditions — Coronary Artery Disease; Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Coronary stent - Tsunami — A coronary angioplasty was done

SUMMARY:
The freedom of choice in medicine is based on the physician's ability to treat their patients with the best available therapy. The armamentarium for percutaneous intervention is frequently determined on the basis of subjective criteria and the experience of the interventional cardiologist. The evaluation of devices used in coronary intervention, especially angiography and its clinical outcomes, has rarely been investigated; the exceptions are studies on stents. Therefore, the freedom of choice for the interventional cardiologist has been challenged, especially because of cost restrictions. This way this study aims to assess the safety and efficacy of a device of a single brand in performing percutaneous transluminal coronary angioplasty (guide catheters, guidewires, balloons, and stents) in selected patients.

ELIGIBILITY:
Inclusion Criteria:

The study included both male and female patients for stent implantation referred for angioplasty of coronary arteries with more than 18 years.

Exclusion Criteria:

* chronic total occlusion angioplasty,
* saphenous graft angioplasty,
* bifurcation angioplasty (lateral branch greater than 1.5 mm)
* plans to perform angioplasty on more than one vessel during the same procedure
* and primary angioplasty in acute myocardial infarction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2011-01; Primary Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Occurrence of: need to change the materials during the procedure (angioplasty). | 12 months